CLINICAL TRIAL: NCT07198269
Title: Comparison of Oxygenation Stability Between Different Ventilators in Mechanically Ventilated Patients During Transport: a Single-blind, Single-center, Parallel-group, Non-inferiority Randomized Controlled Trial
Brief Title: Assessment of A Novel Emergency Transport Ventilator in Mechanically Ventilated Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0931; 2022YFC2403604 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Patients Receiving Invasive Mechanical Ventilation
Keywords: Transport ventilators; Oxygenation stability; Randomized controlled trial; Mechanical ventilation; Non-inferiority

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel high-performance ventilator for transport (Experimental): Mechanically ventilated patients who requiring intra-hospital or inter-hospital transport with various objects will receiving TV80
  Interventions: Device: Intelligent emergency ventilator for transport; Device: high-performance emergency ventilator for transport
- Intelligent ventilator for transport (Active Comparator): Mechanically ventilated patients who requiring intra-hospital or inter-hospital transport with various objects will receiving HAMILTON-T1
  Interventions: Device: Intelligent emergency ventilator for transport; Device: high-performance emergency ventilator for transport

INTERVENTIONS:
Device: Intelligent emergency ventilator for transport — In this study, eligible patients are first evaluated by research staff to confirm that they meet the inclusion criteria. Once eligibility is established, the research team accesses the electronic data capture (EDC) system via a WeChat QR code, where patients are randomly assigned in a 1:1 ratio to either the domestic ventilator group (TV80) or the imported ventilator group (HAMILTON-T1). After randomization, both patient and ventilator preparation procedures are conducted according to a standardized protocol.
Device: high-performance emergency ventilator for transport — In this study, eligible patients are first evaluated by research staff to confirm that they meet the inclusion criteria. Once eligibility is established, the research team accesses the electronic data capture (EDC) system via a WeChat QR code, where patients are randomly assigned in a 1:1 ratio to either the domestic ventilator group (TV80) or the imported ventilator group (HAMILTON-T1). After randomization, both patient and ventilator preparation procedures are conducted according to a standardized protocol.

SUMMARY:
Brief Summary

The goal of this clinical trial is to compare whether the novel high-performance emergency transport ventilator (TV80) differs from the intelligent transport ventilator (HAMILTON-T1) in terms of oxygenation stability when used for transporting mechanically ventilated patients. It will also collect data on the novel ventilator's performance and safety in multiple transport scenarios. The main questions it aims to answer are:

1. Does the novel high-performance emergency transport ventilator (TV80) show non-inferior oxygenation stability (measured by the difference in oxygenation index before and after transport) compared with HAMILTON-T1 in transporting mechanically ventilated patients?
2. What differences exist between the two ventilators in secondary outcomes such as transport preparation time, changes in PaCO2 and pH before and after transport, and variations in tidal volume, FiO2, heart rate, oxygen saturation, and mean arterial pressure?

We will randomly assign eligible mechanically ventilated patients requiring intra-hospital or inter-hospital transport to either TV80 or HAMILTON-T1 group at a 1:1 ratio, and compare the differences in the above outcomes between the two groups.

Participants will:

1. Be screened for eligibility based on inclusion and exclusion criteria, and their legal representatives will sign the informed consent form.
2. Be randomly assigned to use either TV80 or HAMILTON-T1 group during transport.
3. Undergo blood gas analysis 1 hour after airway intervention stabilization (before transport) and within 1 hour after transport completion to calculate the oxygenation index and changes in PaCO2 and pH.
4. Have transport preparation time recorded (from the start of transport preparation, such as suctioning and pipeline organization, to the confirmation of stable vital signs before transport).
5. Have parameters such as tidal volume, FiO2 (recorded by the ventilator) and heart rate, oxygen saturation, mean arterial pressure (monitored by a incorporated module in TV80 or portable monitor along with HAMILTON-T1) recorded during transport to calculate their variations.
6. Be monitored for adverse events during transport; if severe adverse events occur, the trial will be stopped immediately, and appropriate treatment measures will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and < 80 years.
* Patients receiving invasive mechanical ventilation.
* Patients requiring intra-hospital transport or inter-hospital transfer.
* Patients whose legal representatives have provided written informed consent for participation in the trial.

Exclusion Criteria:

* Subjects with shock or hemodynamic instability that has not been treated
* Subjects receiving high-dose vasopressor support (equivalent norepinephrine dose > 1µg/kg/min)
* Patients receiving ECMO support
* Subjects with hemoglobin < 6g/dL
* Subjects with cardiac arrest without resuscitation treatment
* Patients who are moribund or discharged due to deteriorating condition
* Patients with bullae, pneumothorax without closed thoracic drainage, especially tension pneumothorax
* Massive hemoptysis, and respiratory failure caused by massive hemoptysis or severe aspiration
* Pregnant and lactating women
* Patients with mental illness
* Subjects whose legal representatives have not provided informed consent
* Patients without access to trial ventilators during the trial, including when trial ventilators are in use or malfunctioning
* Expected transport duration exceeding 1 hour or combined transport scenarios (helicopter combined with ambulance)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in PaO2/FiO2 before and after transferring | Within 1 hour before and 1 hour after transport
  Arterial blood samples will be collected within 1 hour before and 1 hour after transport. Blood gas analysis will be performed to obtain PaO2 and FiO2 values and calculate the oxygenation index. The difference between the two indices is then determined.

SECONDARY OUTCOMES:
Variation in heart rate before and after transferring | Procedure (From the beginning to the end of transport)
  From the beginning to the end of transport, obtain data recorded manually or from the ventilator to determine the minimum and maximum heart rates during the entire process, and calculate the difference between them
Variation in SPO2 before and after transferring | Within 1 hour before and 1 hour after transport
  From the beginning to the end of transport, retrieve data recorded manually or from the ventilator to identify the minimum and maximum oxygen saturation levels throughout the process, and calculate the difference between them
Variation inPaCO2 before and after transferring | Within 1 hour before and 1 hour after transport
  Arterial blood samples are collected within 1 hour before and 1 hour after transport. Blood gas analysis is performed to obtain PaCO₂ values before and after transport, and the difference between them is calculated
Variation in tidal volume before and after transferring | Within 1 hour before and 1 hour after transport
  From the beginning to the end of transport, retrieve data from the ventilator to identify the minimum and maximum delivered tidal volumes throughout the process, and calculate the difference between them
Difference in pH before and after transferring | Within 1 hour before and 1 hour after transport
  Arterial blood samples are collected within 1 hour before and 1 hour after transport. Blood gas analysis is performed to obtain pH values before and after transport, and the difference between them is calculated.
Variation in FiO2 before and after transferring | Within 1 hour before and 1 hour after transport
  From the beginning to the end of transport, retrieve data from the ventilator to identify the minimum and maximum delivered FiO₂ values throughout the process, and calculate the difference between them
Variation in mean arterial pressure and after transferring | From the beginning to the end of transport
  From the beginning to the end of transport, retrieve data recorded manually or from the ventilator to identify the minimum and maximum mean arterial pressures throughout the process, and calculate the difference between them
Preparing time for transferring | Procedure (The interval from preparing the patient's ventilator and monitor tubing/lines to transferring the patient onto the stretcher)
  The time interval from preparing the patient's ventilator and monitor tubing and lines to transferring the patient onto the stretcher

CONTACTS AND LOCATIONS:
Overall Officials: Shanxiang Xu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cardinale M, Cungi PJ, Bordes J, Cohergne F, Schmitt S, Langlois A, Meaudre E, Lacroix G. Maintaining a high inspired oxygen fraction with the Elisee 350 turbine transport ventilator connected to two portable oxygen concentrators in an austere environment. J Trauma Acute Care Surg. 2020 Sep;89(3):e59-e63. doi: 10.1097/TA.0000000000002792. PMID 32467466
- [Result] Hernandez-Tejedor A, Gonzalez Puebla V, Corral Torres E, Benito Sanchez A, Pinilla Lopez R, Galan Calategui MD. Ventilatory improvement with mechanical ventilator versus bag in non-traumatic out-of-hospital cardiac arrest: SYMEVECA study, phase 1. Resuscitation. 2023 Nov;192:109965. doi: 10.1016/j.resuscitation.2023.109965. Epub 2023 Sep 12. PMID 37709164